CLINICAL TRIAL: NCT01793298
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of ASM-024 Administered by Dry Powder Inhalation to Healthy Subjects and Subjects With Stable Moderate Asthma
Brief Title: Safety, Tolerability and Pharmacokinetics of ASM-024 Administered to Healthy Subjects and Subjects With Moderate Asthma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Asmacure Ltée (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ASM-024/I-II/STA-03
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — ASM-024

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Healthy Subjects - ASM-024 Single Administration (Experimental): Single administration of ascending doses of ASM-024
  Interventions: Drug: ASM-024
- Healthy Subjects - Placebo (Placebo Comparator): Single administration of placebo
- Healthy Subjects - ASM-024 Repeat Administration (Experimental): Repeat administration of ascending doses of ASM-024
  Interventions: Drug: ASM-024
- Healthy Subjects - Placebo Repeat Administration (Placebo Comparator): Repeat administration of ascending doses of placebo
- Subjects with Asthma (Experimental): Repeat administration of ascending doses of ASM-024 or placebo in a crossover fashion
  Interventions: Drug: ASM-024

INTERVENTIONS:
Drug: ASM-024 — Ascending doses of ASM-024
  Arms: Healthy Subjects - ASM-024 Repeat Administration; Healthy Subjects - ASM-024 Single Administration; Subjects with Asthma

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of the dry powder formulation of ASM-024 following single and multiple administration by inhalation of ascending doses in healthy subjects and subjects with stable moderate asthma.

DETAILED DESCRIPTION:
This is a phase I/II, randomized, double-blind, placebo-controlled study of single ascending and multiple ascending doses of ASM-024 administered by dry powder inhalation to healthy subjects and subjects with stable moderate asthma. The goal of this study is to evaluate the safety, tolerability and pharmacokinetic profile of a new, dry powder formulation of ASM-024. The doses that will be tested in subjects with asthma will be determined based on the information collected first in healthy volunteers. In addition to standard safety and tolerability evaluations, the acute effects of the study medication on the airways will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* Healthy male or female adult, 18 to 55 years of age ; non-smoker or former smoker;
* Normal lung function; and
* Normal 12-lead ECG

Asthmatics:

* Male or female adult, 18 to 60 years of age with diagnosis of moderate asthma according to the GINA Guidelines and on regular inhaled corticosteroids with or without short or long-acting beta 2-agonists;
* Non-smoker or former smoker;
* FEV1 ≥ 70 % predicted in the absence of medications for asthma;
* Baseline methacholine PC20 ≤ 16 mg/mL; and
* Normal 12-lead ECG.

Exclusion Criteria:

Healthy Volunteers:

* Clinically significant illness or surgery within 8 weeks prior to first administration of the study medication;
* Significant medical history that, in the Investigator's opinion, may adversely affect participation;
* History of allergy or significant adverse reaction to drugs similar to ASM-024, to nicotine, or to cholinergic drugs or any drugs with a similar chemical structure;
* History of hypersensitivity (anaphylaxis, angioedema) to any drug;
* Use of any drug known to induce or inhibit hepatic drug metabolism, within 30 days prior to first administration of the study medication;
* Positive pregnancy test for female subjects;
* Use of medications known to prolong QT/QTc interval within 14 days prior to the first administration of the study medication;
* Clinically significant 12 lead ECG abnormalities at Screening;;
* Clinically significant physical examination or laboratory findings at Screening;
* History of alcohol or drug abuse;
* Tobacco use within 12 months prior to Screening, or nicotine-containing products within 6 months prior to Screening. History of smoking must be ≤ 10 pack-years;
* Positive hepatitis B or C or HIV test at Screening;
* Investigational drug within 30 days prior to first administration of the study medication, or long-acting investigational drug within 90 days prior to first administration of the study medication;
* Previous exposure to ASM-024; and
* Women of child-bearing potential and male participants unwilling or unable to use accepted methods of birth control.

Asthmatics:

* Clinically significant illness or surgery within 8 weeks prior to first administration of the study medication;
* Significant medical history that, in the Investigator's opinion, may adversely affect participation;
* History of allergy or significant adverse reaction to drugs similar to ASM-024, to nicotine, or to cholinergic drugs or any drugs with a similar chemical structure;
* History of hypersensitivity (anaphylaxis, angioedema) to any drug;
* Use of any drug known to induce or inhibit hepatic drug metabolism, within 30 days prior to first administration of the study medication;
* Positive pregnancy test for female subjects;
* Use of medications known to prolong QT/QTc interval;
* Clinically significant 12 lead ECG at Screening;
* Clinically significant physical examination or laboratory findings or abnormal vital signs;
* Baseline methacholine PC20 > 16 mg/mL at Screening;
* History of illicit drug use or alcohol abuse within 12 months of Screening;
* Tobacco use within 12 months prior to Screening, or nicotine-containing products within 6 months prior to Screening. History of smoking must be ≤ 10 pack-years;
* Positive hepatitis B or C or HIV test at Screening;
* Any of the following concomitant medications preceding the administration of methacholine during Screening and preceding the administration of the study medication at Visit 1: (i) oral or i.v. corticosteroids within 1 month; (ii) inhaled or intranasal corticosteroids within 48 hours; (iii) long-acting beta-2-agonists within 48 hours; (iv) short-acting beta-2-agonists within 8 hours; (v) anticholinergic aerosol within 24 hours; (vi) theophyline-containing products within 48 hours; (vii) NSAIDs within 7 days preceding the administration of methacholine during Screening and throughout the study; and (viii) antihistaminic drugs within 3 days;
* Investigational drug within 30 days of Screening; long-acting investigational drug within 90 days of Screening;
* Previous exposure to ASM-024; and
* Women of child-bearing potential and male participants unwilling or unable to use accepted methods of birth control.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
adverse events, spirometry | up to 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Yvon Cormier, M.D., Study Chair — Asmacure Ltée
Locations (2):
- Canada (2):
  - PharmaNet, Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec